CLINICAL TRIAL: NCT03204799
Title: Metagenomic Analysis of Human Gut Microbiota in Patients With Metabolic Diseases Including Diabetes.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0950
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus; Dyslipidemias
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Metformin; Sodium-Glucose Transporter 2 Inhibitors; Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- normal group: normal group (without diabetes diagnosis/treatment and in normoglycemia
  Interventions: Other: Metformin; Drug: ezetimibe
- prediabetes: high risk, impaired fasting glucose, impaired glucose tolerance
  Interventions: Other: Metformin; Drug: ezetimibe
- drug naive type 2 diabetes: type 2 diabetes, anti-hypoglycemic drug naive
  Interventions: Other: Metformin; Drug: ezetimibe
- type 2 diabetes with metformin monotherapy: type 2 diabetes with metformin monotherapy
  Interventions: Other: Metformin
- type 2 diabetes with SGLT2 inhibitor monotherapy: type 2 diabetes with SGLT2 inhibitor monotherapy
  Interventions: Drug: SGLT2 inhibitor
- dyslipidemia with ezetimibe therapy: dyslipidemia with ezetimibe therapy
  Interventions: Drug: ezetimibe

INTERVENTIONS:
Other: Metformin — newly diagnosed type 2 diabetes patients who start to metformin monotherapy
  Groups: drug naive type 2 diabetes; normal group; prediabetes; type 2 diabetes with metformin monotherapy
Drug: SGLT2 inhibitor — newly diagnosed type 2 diabetes patients who start to SGLT2 inhibitor monotherapy
  Groups: type 2 diabetes with SGLT2 inhibitor monotherapy
Drug: ezetimibe — newly diagnosed dyslipidemia patients who start to ezetimibe therapy
  Groups: drug naive type 2 diabetes; dyslipidemia with ezetimibe therapy; normal group; prediabetes

SUMMARY:
Microbiota is important for immunology, hormonal and metabolic homeostasis in human and could influence on developing diabetes and obesity. Recent studies investigates microbiota by metagenomic sequencing, however, the composite of microbiota and its metabolic role has not been fully determined. Metagenomics and microbiome analysis could early diagnose metabolic disorders and suggest treatment options for metabolic diseases.

In this study, the investigators investigate the composite of microbiota and deduct basic information for treatment models using metagenomic sequencing.

DETAILED DESCRIPTION:
1. Cross-section study: normal/prediabetes/drug naïve type2 diabetes: compare microbiota using metagenomic sequencing among three groups.
2. Observational prospective study: metformin/sodium glucose co-transporter 2 (SGLT2) inhibitor/ezetimibe: compare microbiota using metagenomic sequencing before and after drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* normal group: body mass index [BMI]<23kg/m2, without diabetes mellitus history
* prediabetes group: fasting blood glucose ≥100 mg/dL and <126 mg/dL or postprandial blood glucose ≥140 mg/dL and <200 mg/dL
* type 2 diabetes according to ADA(American Diabetes Association) guideline (1) fasting blood glucose ≥126 mg/dL, (2) random blood glucose ≥200 mg/dL and with typical diabetes symptoms, (3) glycated hemoglobin A1c ≥6.5% and anti-hypoglycemic drug naive
* patients with type 2 diabetes, metformin monotherapy, SGLT2 inhibitor monotherapy
* patients with dyslipidemia, ezetimibe therapy

Exclusion Criteria:

* inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* history of stomach, small intestine or colon resection operation
* on antibiotics therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes patients with oral hypoglycemic agent/insulin naive
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-12-17 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12-16 (Estimated)

PRIMARY OUTCOMES:
Metagenomic profile change | 10 days (acute effect)
  Stool metagenomic profile change in acute and chronic phase
Metagenomic profile change | 3 months (chronic effect)
  Stool metagenomic profile change in acute and chronic phase

SECONDARY OUTCOMES:
blood glucose change | 3 months
  fasting blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of Internal Medicine, Division of Endocrinology, Severance Hospital, Diabetes center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No